CLINICAL TRIAL: NCT00170976
Title: A 54 Week, Extension to the Double-blind, Multicenter, Multifactorial, Placebo-controlled, Study to Evaluate the Efficacy and Safety of Valsartan (160 mg and 320 mg) and Amlodipine (10 mg) Combined and Alone in Hypertensive Patients
Brief Title: A Year Long Study to Evaluate the Safety of the Combination of Valsartan (320 mg) and Amlodipine (5 mg) in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489A2307E1
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: HYPERTENSION
Keywords: HYPERTENSION, VALSARTAN, AMLODIPINE< SAFETY
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan + amlodipine

SUMMARY:
A ONE YEAR SAFETY STUDY FOR PATIENTS WHO COMPLETE STUDY VAA489A2307.

ELIGIBILITY:
Inclusion Criteria:

* SUCCESSFUL COMPLETION OF VAA489A2307 CORE TRIAL
* VISIT 7 BLOOD PRESSURE MUST BE MSDBP ≤ 95 mmHg AND MSSBP ≤ 150 mmHg

Exclusion Criteria:

* PATIENTS WHO EXPERIENCED ANY ADVERSE EVENTS CONSIDERED SERIOUS AND DRUG RELATED IN VAA489A2307 CORE

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events at each study visit for 6 or 12 months

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure from baseline after 6 or 12 months
Change from baseline in systolic blood pressure from baseline after 6 or 12 months
Change from baseline in standing diastolic and systolic blood pressure after 6 or 12 months
Change from baseline in sitting and standing pulse after 6 or 12 months
Hematology and blood chemistry after 6 or 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Sites in germany, Multiple Locations, Germany
- Novartis Pharmaceuticals, Basel, Switzerland